CLINICAL TRIAL: NCT07048483
Title: REEL DIETS: Researching Engagement With Educational Lifestyle Content: a Diet-based Intervention for Eating and Self-efficacy
Brief Title: Researching Engagement With Educational Lifestyle Content
Acronym: REEL DIETS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Enid Keseko, Principal Investigator, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00145670
Record Dates: First submitted 2025-06-23; First posted 2025-07-02 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Diet Quality
Keywords: health messaging; self-efficacy for healthy eating; diet quality; overweight/obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Nutrition Assessment; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audio-visual messaging (Experimental): Participants will watch audio-visual messages on healthy eating per week for four weeks, presented through videos and films.
  Interventions: Behavioral: Nutrition Education
- Handouts (Active Comparator): Participants will not engage with any audio-visual messages but will receive educational materials about healthy eating in the form of handouts.
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: Nutrition Education — This intervention uses curated audio-visual messages through videos and films to engage participants in learning about healthy eating behaviors, followed by structured, brief discussions designed to reflect on the content and relate it to personal dietary habits. The intervention leverages narrative-based media to increase self-efficacy for healthy eating.
  Arms: Audio-visual messaging
Other: control group — Educational materials about food and healthy in the form of handouts will be provided to participants to review.
  Arms: Handouts

SUMMARY:
The goal of this study is to examine how different types of health messages affect people's self efficacy for healthy eating and diet quality. Eligible adult participants with overweight/obesity will be randomized into one of two groups: the intervention group, which will engage with audio-visual messages per week for four weeks, or the control group, which will not engage with any audio-visual messages but will receive written educational materials about healthy eating per week for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* BMI of ≥25 kg/m²
* Have no dietary restrictions
* Have access to the internet
* Have a Netflix subscription
* Have availability to engage in group discussions

Exclusion Criteria:

* Currently following a vegan or vegetarian diet
* Have a diagnosis of an eating disorder
* Pregnant or breastfeeding
* Have recent participation in a weight loss or nutrition intervention (within the past 6 months)
* Have any medical condition requiring a medically prescribed diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2025-07-07 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Diet quality | 4 weeks
  Rapid Eating Assessment for Participants - Short form survey. Total scores range from 13 to 39. Higher scores indicate better diet quality.
Self-efficacy | 4 weeks
  Healthy Eating and Weight Self-Efficacy scale. Total scores range from 11 to 55. Higher scores indicate greater self-efficacy for healthy eating and weight control behaviors.
Self-efficacy | 4 weeks
  Fruit and Vegetable Intake Self Efficacy scale. Score range is 1 to 7 (per item); mean scores calculated across 22 items. Higher scores indicate greater self-efficacy in consuming fruits or vegetables.

SECONDARY OUTCOMES:
Intentions | 4 weeks
  Intentions to eat healthy scale. Each item is rated on a 7-point bipolar scale, with response options ranging from -3 to +3, where higher scores indicate stronger intentions to adopt a healthy diet.

CONTACTS AND LOCATIONS:
Locations (1):
- Online., Columbia, South Carolina, United States